CLINICAL TRIAL: NCT05544513
Title: Effects of Oral Iron Supplementation on Gut Microbiota in Patients With Chronic Kidney Disease
Brief Title: Oral Iron Supplementation for Patients With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DeniseMafra14
Record Dates: First submitted 2022-01-04; First posted 2022-09-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Renal Disease; Iron-Deficiency Anemia; Anemia of Chronic Kidney Disease; Dysbiosis
Keywords: hepcidin; inflammation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency; Dysbiosis; Inflammation | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (Experimental): participants will receive one ferrous sulfate capsule (120 mg of elemental iron) on Mondays, Wednesdays and Fridays
  Interventions: Drug: Ferrous sulfate 3 days week
- Group II (Active Comparator): participants will receive one ferrous sulfate (120 mg of elemental iron) capsule daily (except on Sundays)
  Interventions: Drug: Ferrous sulfate daily
- Group III (Active Comparator): participants will receive one ferrous sulfate capsule (240mg of elemental iron) on Mondays, Wednesdays and fridays
  Interventions: Drug: Ferrous sulfate higher concentration

INTERVENTIONS:
Drug: Ferrous sulfate 3 days week — Participants will receive one ferrous sulfate capsule (120 mg of elemental iron) on Mondays, Wednesdays and Fridays
  Arms: Group I
Drug: Ferrous sulfate daily — Participants will receive one ferrous sulfate (120 mg of elemental iron) capsule daily (except on Sundays)
  Arms: Group II
Drug: Ferrous sulfate higher concentration — Participants will receive one ferrous sulfate capsule (240mg of elemental iron) on Mondays, Wednesdays and fridays
  Arms: Group III

SUMMARY:
The hypothesis of this research is that oral iron prescribed in a single dose in alternate day could mitigate the side effects with regard to intestinal microbiota, inflammation, oxidative stress and improve the hematological profile when compared to daily oral iron prescription

DETAILED DESCRIPTION:
chronic kidney disease triggers several changes in the body, anemia is one of the first disorders that appear in chronic kidney disease patients. The anemia in this patient is multifactorial, the main cause being relative erythropoietin deficiency, although iron deficiency is also common. In this context, the need for oral iron supplementation is a way of both treating iron deficiency and optimizing the use of agents that stimulate erythropoiesis. However, this replacement can cause iron overload, increasing the production of reactive oxygen species and, consequently, oxidative stress, and also alter the intestinal microbiota leading to poor iron absorption, worsening the prognosis of chronic kidney disease. The current routine for iron supplementation for these patients is to offer oral iron daily, which can be more harmful than when given on alternate days. However, there are few studies comparing the two prescriptions.

In this context, since no study to date has been carried out to show the aforementioned effects in the participant with chronic kidney disease, this randomized clinical trial aims to assess the effects of daily or alternate-day oral iron supplementation on gut microbiota composition in participants with chronic kidney disease (glomerular filtration rate (GFR) below 30 mL/min) for 3 months. The project will also compare the effects of both prescriptions on serum hepcidin levels, markers of oxidative stress and inflammation, and on routine hematological and biochemical parameters.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 to 75 years Clinical diagnosis of Chronic Kidney Disease Conservative treatment group: chronic kidney disease stages 3 and 5

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Autoimmune diseases
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-12-29 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in cytokines plasma levels measured by ELISA after supplementation with oral iron | 2 months
  cytokines plasma levels

SECONDARY OUTCOMES:
Change in uremic toxin plasma levels after supplementation with oral iron | 2 months
  Get blood samples to evaluate the supplementation effects in uremic toxins such as indoxyl sulfate, p-cresyl sulfate

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil